CLINICAL TRIAL: NCT05468229
Title: Effects of Dorzagliatin on 1st Phase Insulin and Beta-cell Glucose Sensitivity in Individuals With Impaired and Normal Glucose Tolerance
Brief Title: Dorzagliatin and 1st Phase Insulin and Beta-cell Glucose Sensitivity in IGT and NGT
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Juliana Chan, Professor, Chinese University of Hong Kong
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Treatment
Other Study IDs: 2021.516-T
Record Dates: First submitted 2022-07-19; First posted 2022-07-21 (Actual); Last update posted 2022-07-25 (Actual); Status verified 2022-07

CONDITIONS: Glucose Intolerance
MeSH Terms: conditions — Glucose Intolerance | interventions — Dorzagliatin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Masking Description: double blind placebo controlled
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- dorzagliatin (Active Comparator): Dorzagliatin 50 mg single dose
  Interventions: Drug: Dorzagliatin
- placebo (Placebo Comparator): matching placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dorzagliatin — single oral dose of dorzagliatin 50 mg
  Arms: dorzagliatin
Drug: Placebo — Matching placebo
  Arms: placebo

SUMMARY:
Dorzagliatin, a novel dual allosteric activator of glucokinase. reduces blood glucose by increasing insulin secretion by enhancing sensitivity of beta cells to glucose. In this placebo controlled cross over study, we examined the effects of dorzagliatin in people with impaired glucose tolerance and normal glucose tolerance.

DETAILED DESCRIPTION:
Objective

To investigate the acute effects of a single dose dorzagliatin on first phase insulin secretion and beta cell glucose sensitivity (βCGS) in individuals with impaired and normal glucose tolerance

Methodology and rationale:

A total of 20 subjects will be recruited, 10 in impaired glucose tolerant (IGT) and 10 in normal glucose tolerant (NGT) groups, respectively. Eligible participants will have a two-hour hyperglycemic clamp following a single dose of dorzagliatin or placebo in a randomized crossover fashion on V2 or V3. Subjects will be randomized to dorzagliatin 50mg or placebo in the IGT and NGT groups. Arterialized blood glucose (venous blood drawn from back of the hand placed in a temperature regulated box), measured every 5 minutes at the bedside Yellow Spring Instrument (YSI) or EKF glucose analyser, will be maintained at 12 mmol/l using an infusion of dextrose. Blood will be sampled for insulin and C-peptide at regular intervals for evaluation of first and second phase insulin secretion. Glucagon-like peptide-1 (GLP-1) and glucagon will be evaluated at regular intervals during the clamp studies. After 14 ± 2 days washout out (Day 14), participants will receive a single dose of dorzagliatin or matched placebo followed by a repeat hyperglycemic clamp to evaluate differences in beta-cell function.

ELIGIBILITY:
Inclusion Criteria:

1. Individuals aged ≥ 18 years but < 65years
2. Male or female
3. Body mass index of over 18 kg/m2 and < 30 kg/m2

Additional inclusion criteria for IGT group

* Fasting plasma glucose <7.0 mmol/L and HbA1c < 6.5%
* 2 hour plasma glucose ≥7.8 and <11.1 mmol/L on 75g oral glucose tolerance test (OGTT)
* Never been treated with glucose lowering drugs (including traditional Chinese medicine for glycemic control)

Additional inclusion criteria for NGT group

* Fasting plasma glucose <5.6 mmol/L and HbA1c < 5.7%
* 2 hour plasma glucose <7.8 mmol/L on 75g oral glucose tolerance test (OGTT)
* Never been treated with glucose lowering drugs (including traditional Chinese medicine for glycemic control

Exclusion Criteria:

1. Subjects who do not agree to participate in this study.
2. Country of birth is unknown.
3. Body weight less than 45kg.
4. Acute phase of cerebrovascular and cardiovascular diseases (within 6 months of recruitment).
5. Subjects with severe renal dysfunction as defined by eGFR <30 ml/min/1.73m2 or patients receiving renal dialysis (such as haemodialysis or continuous ambulatory peritoneal dialysis).
6. Severe hepatic dysfunction as defined by AST and/or ALT > 3 times upper limit of normal.
7. Severe cardiovascular disease, history of stroke, heart failure (NYHA III or IV) or history of myocardial infarction within last 12 months.
8. History of drug abuse or excessive alcohol intake based on investigator judgment.
9. History of diabetes mellitus.
10. Dehydration, diarrhoea or vomiting at the time of recruitment.
11. Subjects with severe infection, in perioperative period or with serious injury at the time of recruitment.
12. Subjects with anaemia (Haemoglobin <11.0mg/dL or haematocrit <0.35 ) at screening, known iron deficiency, haemoglobinopathies or anaemia due to chronic disease.
13. Pregnant or lactating or intending to become pregnant within 30 days after last dose of study drug.
14. Participation in a clinical trial with investigational product within 30 days before enrolment.
15. Donation or loss of blood (excluding the volume of blood that will be drawn during screening procedures) as follows: ≥300 mL of blood within 30 days prior to study drug administration.
16. Subjects judged unsuitable for the study based on investigator judgment.
17. Use of strong or moderate CYP3A4 inhibitors or inducers and cannot be discontinued.
18. Unwilling or unable to follow protocol requirements

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 20 (Estimated)
Dates: Start 2022-08 (Estimated); Primary Completion 2023-04 (Estimated); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
2-hour hyperglycemic clamp | 2-hour
  first phase insulin secretion

IPD SHARING:
Plan to Share IPD: No